CLINICAL TRIAL: NCT06467591
Title: Prediction of Long-term Survival and Chemotherapy Benefit in Elderly Advanced Gastric Cancer Patients Based on the mCNS Model of Nutritional Control State Score and Sarcopenia.
Brief Title: Prediction Model for Advanced Gastric Cancer in Elderly
Status: Completed | Type: Observational
Sponsor: Chang-Ming Huang, Prof. (Other)
Responsible Party: Sponsor-Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: 2024KY076
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Stomach Neoplasms; Aged
Keywords: Stomach Neoplasms; Prognosis; Elderly; Prediction Model
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop and validate a Nomogram (mCNS) model for predicting long-term survival in elderly patients following curative resection for advanced gastric cancer. The study is a retrospective multi-center analysis involving 924 gastric cancer patients treated at the Department of Gastrointestinal Surgery of the Affiliated Union Hospital of Fujian Medical University between 2009 and 2013, and 512 patients aged 65 and above who underwent gastric resection at the Affiliated Zhongshan Hospital of Dalian University between 2011 and 2018. An online prognostic tool is introduced to assist clinicians in predicting patient prognosis and customizing treatment and follow-up strategies.

DETAILED DESCRIPTION:
Data were collected from 1436 gastric cancer patients, of which 555 elderly patients with advanced gastric cancer were ultimately included after applying exclusion criteria. Patients were divided into training and testing cohorts from the Fujian Medical University Affiliated Union Hospital and Dalian University Affiliated Zhongshan Hospital. The study was approved by the institutional review boards with a waiver of informed consent due to the use of anonymized secondary data. The analysis utilized the Cox proportional hazards model to select key variables for predicting overall survival (OS). The study also implemented rigorous data handling procedures, including multiple imputations for missing data. The development of an online prognostic tool based on the Nomogram model is part of the project, designed to provide real-time survival predictions through a user-friendly interface for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed as primary gastric adenocarcinoma by preoperative gastric endoscopy pathology;
* Underwent R0 laparoscopic radical gastrectomy for gastric cancer;
* Pathological stage T2-4a-N+;
* Age ≥ 65 years.

Exclusion Criteria:

* Pathological stage T1 and T2N0;
* Age < 65 years;
* Presence of peritoneal or distant metastasis confirmed before or during surgery;
* Received neoadjuvant chemotherapy before surgery;
* Remnant gastric cancer;
* Emergency surgery or palliative exploratory surgery;
* Preoperative abdominal CT scan not available or preoperative examination time > 1 month;
* Survival time less than 1 month;
* Incomplete clinical and pathological data.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population comprises elderly patients, aged 65 and above, diagnosed with gastric cancer and who underwent curative gastrectomy within a ten-year period from January 2009 to December 2018. Participants were selected from two major tertiary care centers in China, ensuring a comprehensive representation of the demographic. Strict adherence to selection criteria ensured the use of a consistent and high-quality dataset for subsequent analysis in developing a robust prognostic model. The study focuses on the elderly demographic, addressing a significant gap in prognostic tools for this age group, which often presents with distinct clinical and therapeutic challenges.
Sampling Method: Non-Probability Sample
Enrollment: 1436 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
5-Year Overall Survival | 5 years or 60 months.
  The proportion of patients who are alive at five years after treatment for elderly gastric cancer patients.

SECONDARY OUTCOMES:
3-Year Overall Survival | 3 years or 36 months.
  The proportion of patients who have survived without any signs or symptoms of gastric cancer for 3 years after the initial treatment.
1-Year Overall Survival | 1 years or 12 months.
  The proportion of patients who have survived without any signs or symptoms of gastric cancer for 1 years after the initial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, M.D, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Department of Gastric Surgery， Fujian Medical University Union Hospital, Fuzhou, Fujian, China